CLINICAL TRIAL: NCT00049556
Title: Phase II Pilot Study of Clinical Activity and Proteomic Pathway Profiling of the EGFR Inhibitor, ZD1839 (Iressa; Gefitinib), in Patients With Epithelial Ovarian Cancer or Cervical Cancer
Brief Title: Gefitinib in Treating Patients With Cervical Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000258117; NCI-02-C-0303; NCI-5561; NCT00046007 (obsolete NCT alias)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2006-01

CONDITIONS: Cervical Cancer; Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: fallopian tube cancer; borderline ovarian surface epithelial-stromal tumor; primary peritoneal cavity cancer; recurrent cervical cancer; recurrent ovarian epithelial cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Gefitinib; Immunohistochemistry; Spectrometry, Mass, Matrix-Assisted Laser Desorption-Ionization; Biopsy; Sentinel Lymph Node Biopsy

INTERVENTIONS:
Drug: gefitinib
Other: immunohistochemistry staining method
Other: surface-enhanced laser desorption/ionization-time of flight mass spectrometry
Procedure: biopsy
Procedure: sentinel lymph node biopsy

SUMMARY:
RATIONALE: Biological therapies such as gefitinib may interfere with the growth of the tumor cells and slow the growth of cervical cancer. Comparing results of diagnostic procedures performed before, during, and after treatment with gefitinib may help doctors predict a patient's response to treatment and help plan the most effective treatment.

PURPOSE: This phase II trial is studying how well gefitinib works in treating patients with cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the reduction in phosphorylation of epidermal growth factor receptor (EGFR), AKT, and ERK by proteomics in tumor and normal skin of patients with ovarian epithelial cancer or cervical cancer receiving gefitinib. (Open to accrual for cervical cancer patients only as of 4/5/2005)
* Determine the clinical activity of this drug in these patients.
* Determine the toxicity of this drug in these patients.
* Correlate the biologic modulation of EGFR, ERK, and AKT by this drug with outcome and toxic effects in these patients.
* Correlate EGFR modulation in skin with outcome and toxic effects in patients treated with this drug.
* Correlate expression of EGFR and phosphorylated-EGFR in tissue biopsies from these patients with biochemical modulation and outcome.
* Determine the application of surface-enhanced laser desorption and ionization with time-of-flight detection (SELDI-TOF) and artificial intelligence bioinformatics to serially obtained serum samples for predicting response and toxic effects in these patients.

OUTLINE: Patients are stratified according to disease (cervical cancer vs ovarian epithelial, fallopian tube, and primary peritoneal cancer). (Open to accrual for cervical cancer patients only as of 4/5/2005)

Patients receive oral gefitinib daily. Treatment continues every 28 days in the absence of disease progression or unacceptable toxicity.

Biopsies of a sentinel lesion (with CT guidance or laparoscopy) are obtained at baseline and at 4 weeks. Skin biopsies of unaffected areas are also obtained at these time points. Tissue is examined using immunohistochemical methods. Proteomic profiling using surface-enhanced laser desorption/ionization with time-of-flight (SELDI-TOF) mass spectrometry is conducted on serum at baseline and then every 4 weeks.

Patients are followed monthly.

PROJECTED ACCRUAL: A total of 30-40 patients (15-20 per stratum) will be accrued for this study within 10-12 months. (Open to accrual for cervical cancer patients only as of 4/5/2005)

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial cancer or cervical cancer (open to accrual for cervical cancer patients only as of 4/5/2005)

  * Relapsed or refractory
* The following are also eligible: (open to accrual for cervical cancer patients only as of 4/5/2005)

  * Cancer of the fallopian tube
  * Primary peritoneal cancer
  * Cancer with low malignant potential and an invasive recurrence
* Block or recuts of primary tumor or recent resection specimen of a metastatic site required
* Measurable disease with a sentinel lesion adequate for core biopsy by percutaneous biopsy or laparoscopy
* No CNS involvement

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC greater than 3,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic

* Bilirubin less than 1.5 mg/dL
* AST and ALT no greater than 2.5 times upper limit of normal

Renal

* Creatinine less than 1.5 mg/dL

Cardiovascular

* No myocardial infarction within the past 6 months
* No unstable dysrhythmia within the past 6 months

Other

* No other invasive malignancy within the past 5 years except noninvasive nonmelanoma skin cancer
* No active ocular inflammation or infection
* No active infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior cetuximab or monoclonal antibody ABX-EGF

Chemotherapy

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered

Endocrine therapy

* At least 4 weeks since prior hormonal therapy and recovered
* No concurrent tamoxifen

Radiotherapy

* At least 4 weeks since prior radiotherapy and recovered

Surgery

* Recovered from prior oncologic or other major surgery

Other

* No prior epidermal growth factor receptor inhibitory agents (e.g., OSI-774)
* No concurrent antiretroviral therapy
* No concurrent itraconozole, ketoconazole, erythromycin, verapamil, chlorpromazine, amiodarone, or chloroquine
* No concurrent drugs known to induce CYP3A4 enzymes (e.g., phenytoin, carbamazepine, rifampicin, barbiturates, oxacarbazepine, rifapentine, or Hypericum perforatum)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Biochem. modulation of EGFR signal transduction pathways in tumor by tissue lysate array reduction in phosphorylation of EGFR , AKT, and ERK in tumor biopsies at baseline and at 4 weeks during therapy

SECONDARY OUTCOMES:
Biochem. modulation of EGFR signal transduction pathways in skin biopsy tissue by tissue lysate array reduction in phosphorylation of EGFR , AKT, and ERK in skin biopsies at baseline and at 4 weeks during therapy
Clinical activity of gefitinib as measured by CT scan of chest/abdomen/pelvis every 8 weeks
Toxicity as measured by laboratory testing, history, physical exam, and patient diary every 4 weeks
Skin as a surrogate site for study of EGFR modulation and correlation with outcome and toxicity as measured by tissue lysate arrays at baseline and 4 weeks after the start of study therapy
Potential collateral activation of other signal pathways in tumor and skin as measured by tissue lysate arrays at baseline and 4 weeks after the start of study therapy
Expression of EGFR and phosphorylated-EGFR (pY-EGFR) as measured by tissue lysate arrays at baseline and 4 weeks after the start of study therapy
Prediction of response and/or toxicity by serially obtained serum samples using surface-enhanced laser desorption and ionization with time-of-flight detection (SELDI-TOF) and artificial intelligence bioinformatics at baseline and then monthly

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Kwitkowski, MS, RN, CS, CRNP, Study Chair — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland

REFERENCES:
- [Result] Posadas EM, Liel MS, Kwitkowski V, Minasian L, Godwin AK, Hussain MM, Espina V, Wood BJ, Steinberg SM, Kohn EC. A phase II and pharmacodynamic study of gefitinib in patients with refractory or recurrent epithelial ovarian cancer. Cancer. 2007 Apr 1;109(7):1323-30. doi: 10.1002/cncr.22545. PMID 17330838
- [Result] Liel MS, Espina V, Pazzagli C, et al.: Phase II study of gefitinib in epithelial ovarian cancer: Proteomic pathway profiling in tumor biopsies. [Abstract] American Association for Cancer Research: 96th Annual Meeting, April 16-20, 2005, Anaheim/Orange County, CA. A-5745, 2005. .